CLINICAL TRIAL: NCT01177501
Title: Phase I Trial of High-dose Topotecan in Association With Carboplatin, With Peripheral Blood Stem Cell Support in Patients With First Relapsed Ovarian Carcinoma Without Platinum-treatment Since 6-12 Months
Brief Title: Trial of High Dose Topotecan With Carboplatin in Patients With Relapsed Ovarian Carcinoma
Acronym: ITOV04
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: choice of the principal investigator
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 050603
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Ovarian Cancer; Relapses
Keywords: Ovarian cancer; Topotecan; Carboplatine; Higt dose chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topotecan (Experimental)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — Six sequential doses established in the absence of limiting toxicity, as follows : 7.5 - 8.0 - 8.5 - 9.0 - 10.0 mg/m²

SUMMARY:
The early relapse of ovarian cancer occurring within 6 months of chemotherapy including platinum regimen are called relapses 'platinum resistant' consecutively patients die quickly of their disease. For relapses occurring between 6 and 12 months, no recommendation occur and few studies are conducted. Therefore it seems interesting to develop a research on intensive chemotherapy using a combination of carboplatin (a drug widely used in most ovarian cancer) with Topotecan , use in a high dose protocol. Topotecan has demonstrated its efficacy in relapse ovarian cancer and its possible use in high doses, a recent study (ITOV01) have demonstrated the feasibility of dose escalation of topotecan monotherapy (MTD set at 9 mg / m² / dx 5 days). This project is a feasibility research of the combination of topotecan and carboplatin in a high dose escalation protocol for early ovarian cancer relapse occurring 6 to 12 months after conventional chemotherapy-based platinum salts.

DETAILED DESCRIPTION:
The combination Topotecan plus carboplatin at high doses has been published by Miles Prince et al in 2001. In a triple combination, the authors were able to define the Maximum Tolerated Dose (MTD) of 3.5 mg / m² / day x 5 days for topotecan, 250 mg / m² for paclitaxel and AUC at 12 for carboplatin (46). The MTD of topotecan combined with carboplatin (AUC 16) and VP 16 could not be determined by Carroll et al (47). However, in the study ITOV01bis (ASCO abstract 2007 No. 1661), the MTD of topotecan was determined in combination with cyclophosphamide at 120 mg / kg and was fixed at 9 mg/m2/jx 5 days, the same as the DMT used in monotherapy ITOV 01).

Studies related above, the combination of high dose of topotecan and carboplatin seems possible with a limited dose of carboplatin at AUC 20, an allocation of 5 days for both drugs [with a fixed daily AUC 4 for carboplatin , same as the program TAXIF I in germ cell tumors, published by our team (Annual Oncology 2004) as well as TAXIF II developed by Tenon's hospital] with an administration time of 30 minutes daily for topotecan and 2 hours for carboplatin.

these data justify the pattern of our study:

* established treatment of 5 consecutive days provides the best therapeutic index,
* infusion of 30 minutes, seems to give less non-haematological toxicity compare to continuous infusion, which prevailed in the trial ITOV 01,
* Rescue by blood stem cells (collected by chemotherapy mobilization-type high-dose cyclophosphamide followed by hematopoietic growth factors (G-CSF, Filgrastim) reinjection is scheduled to H96 after the treatment end ,
* six sequential doses established in the absence of limiting toxicity, as follows: 7.5 - 8.0 - 8.5 - 9.0 - 9.5 - 10.0 mg/m2. Steps 9.5 mg / m² and 10 mg / m will be discussed after approval by an independent committee in charge of the studyContinuation of Topotecan at conventional dose can be done thanks to clinical data based on efficacy and tolerance

ELIGIBILITY:
Inclusion Criteria:

* Primary ovarian or tubal adenocarcinoma, or peritoneal carcinoma histologically proved
* Age between 18 and 65
* ECOG criteria £ 2
* Patients with first relapsed ovarian carcinoma without platinum-treatment since 6-12 months and after first-line therapy with platinum salt and taxanes together or successively
* Negative viral serology (HbS, HbC and HIV)
* Informed consent
* Patients with social security

Exclusion Criteria:

* Refractory (relapse < 6 months) or sensitive (relapse > 12 months) relapsed ovarian carcinoma
* Life expectancy < 3 months
* Previous treatment with pelvic radiography
* Previous treatment with Topotecan or other topoisomer I inhibitor
* Non resolutive intestinal obstruction under symptomatic treatment
* Creatinine > or equal at 1.25N and/or creatinine clearance < or equal at 60 ml/mn
* Bilirubin > 1.25N ; transaminase and alkaline phosphatase > 2N (3N if hepatic metastases were present)
* Abnormal heart (ultrasound only) (FR < 30%; FEVG < 50%)
* White blood cells < or equal at 4.0 x 109/L, Neutrophils < or equal at 1.5 x 109/L, platelets < or equal at 100 x 109/L
* Neuropathy: grade > or equal at 2
* Epilepsy
* Symptomatic cerebral metastases
* Serious psychiatric pathology
* Uncontrolled serious infection
* Patient that already received peripheral blood stem cell support
* Haematopoeitic growth factors allergy
* More than one line chemotherapy
* Impossibility to use an central veinous access
* Hypersensibility to carboplatin or other platinum containing products
* Participation to an other clinical trial
* Absence of effective contraception

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Identification of the maximum tolerated dose (MTD) of topotecan at 6 weeks | at 6 weeks after the first administration of topotecan
  Evaluation of limiting toxicities (toxic death, grade IV non-hematopoietic or haematopoietic toxicity)of topotecan

SECONDARY OUTCOMES:
Pharmacokinetic of topotecan | At 1 and 5 days after the first administration of topotecan
Pharmacokinetic of carboplatin | At 1 and 5 days after the first administration of topotecan
The response to therapy | From the first day of the administration of topotecan to 2 years
The duration of response and the overall survival | From the first day of the administration of topotecan to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Selle, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Frédéric Selle, Paris, France

REFERENCES:
- [Background] McGuire WP, Hoskins WJ, Brady MF, Kucera PR, Partridge EE, Look KY, Clarke-Pearson DL, Davidson M. Cyclophosphamide and cisplatin versus paclitaxel and cisplatin: a phase III randomized trial in patients with suboptimal stage III/IV ovarian cancer (from the Gynecologic Oncology Group). Semin Oncol. 1996 Oct;23(5 Suppl 12):40-7. PMID 8941409
- [Background] Trimble EL, Adams JD, Vena D, Hawkins MJ, Friedman MA, Fisherman JS, Christian MC, Canetta R, Onetto N, Hayn R, et al. Paclitaxel for platinum-refractory ovarian cancer: results from the first 1,000 patients registered to National Cancer Institute Treatment Referral Center 9103. J Clin Oncol. 1993 Dec;11(12):2405-10. doi: 10.1200/JCO.1993.11.12.2405. PMID 7902426
- [Background] Lotz JP, Bouleuc C, Andre T, Touboul E, Macovei C, Hannoun L, Lefranc JP, Houry S, Uzan S, Izrael V. Tandem high-dose chemotherapy with ifosfamide, carboplatin, and teniposide with autologous bone marrow transplantation for the treatment of poor prognosis common epithelial ovarian carcinoma. Cancer. 1996 Jun 15;77(12):2550-9. doi: 10.1002/(SICI)1097-0142(19960615)77:123.0.CO;2-R. PMID 8640705
- [Background] Mulder PO, Willemse PH, Aalders JG, de Vries EG, Sleijfer DT, Sibinga CT, Mulder NH. High-dose chemotherapy with autologous bone marrow transplantation in patients with refractory ovarian cancer. Eur J Cancer Clin Oncol. 1989 Apr;25(4):645-9. doi: 10.1016/0277-5379(89)90199-5. PMID 2653845
- [Background] Dauplat J, Legros M, Condat P, Ferriere JP, Ben Ahmed S, Plagne R. High-dose melphalan and autologous bone marrow support for treatment of ovarian carcinoma with positive second-look operation. Gynecol Oncol. 1989 Sep;34(3):294-8. doi: 10.1016/0090-8258(89)90161-3. PMID 2670694
- [Background] Viens P, Maraninchi D, Legros M, Oberling F, Philip T, Herve P, Plagne R, Dufour P, Bergerat JP, Guastalla JP, et al. High dose melphalan and autologous marrow rescue in advanced epithelial ovarian carcinomas: a retrospective analysis of 35 patients treated in France. Bone Marrow Transplant. 1990 Apr;5(4):227-33. PMID 2337735
- [Background] Shpall EJ, Clarke-Pearson D, Soper JT, Berchuck A, Jones RB, Bast RC Jr, Ross M, Lidor Y, Vanacek K, Tyler T, et al. High-dose alkylating agent chemotherapy with autologous bone marrow support in patients with stage III/IV epithelial ovarian cancer. Gynecol Oncol. 1990 Sep;38(3):386-91. doi: 10.1016/0090-8258(90)90079-z. No abstract available. PMID 2121627
- [Background] Broun ER, Belinson JL, Berek JS, McIntosh D, Hurd D, Ball H, Williams S. Salvage therapy for recurrent and refractory ovarian cancer with high-dose chemotherapy and autologous bone marrow support: a Gynecologic Oncology Group pilot study. Gynecol Oncol. 1994 Aug;54(2):142-6. doi: 10.1006/gyno.1994.1183. PMID 8063237
- [Background] Murakami M, Shinozuka T, Kuroshima Y, Tokuda Y, Tajima T. High-dose chemotherapy with autologous bone marrow transplantation for the treatment of malignant ovarian tumors. Semin Oncol. 1994 Feb;21(1 Suppl 1):29-32. No abstract available. PMID 8153654
- [Background] Stiff PJ, McKenzie RS, Alberts DS, Sosman JA, Dolan JR, Rad N, McCloskey T. Phase I clinical and pharmacokinetic study of high-dose mitoxantrone combined with carboplatin, cyclophosphamide, and autologous bone marrow rescue: high response rate for refractory ovarian carcinoma. J Clin Oncol. 1994 Jan;12(1):176-83. doi: 10.1200/JCO.1994.12.1.176. PMID 8270975
- [Background] Legros M, Dauplat J, Fleury J, Cure H, Suzanne F, Chassagne J, Bay JO, Sol C, Canis M, Condat P, Choufi B, Tavernier F, Glenat C, Chollet P, Plagne R. High-dose chemotherapy with hematopoietic rescue in patients with stage III to IV ovarian cancer: long-term results. J Clin Oncol. 1997 Apr;15(4):1302-8. doi: 10.1200/JCO.1997.15.4.1302. PMID 9193321
- [Background] Stiff PJ, Bayer R, Kerger C, Potkul RK, Malhotra D, Peace DJ, Smith D, Fisher SG. High-dose chemotherapy with autologous transplantation for persistent/relapsed ovarian cancer: a multivariate analysis of survival for 100 consecutively treated patients. J Clin Oncol. 1997 Apr;15(4):1309-17. doi: 10.1200/JCO.1997.15.4.1309. PMID 9193322
- [Background] Ledermann JA, Herd R, Maraninchi D, Viens P, Buclon M, Philip T, Cure H, Lotz JP, Chauvin F, Ferrante P, Rosti G. High-dose chemotherapy for ovarian carcinoma: long-term results from the Solid Tumour Registry of the European Group for Blood and Marrow Transplantation (EBMT). Ann Oncol. 2001 May;12(5):693-9. doi: 10.1023/a:1011136807190. PMID 11432630
- [Background] Rowinsky EK, Grochow LB, Hendricks CB, Ettinger DS, Forastiere AA, Hurowitz LA, McGuire WP, Sartorius SE, Lubejko BG, Kaufmann SH, et al. Phase I and pharmacologic study of topotecan: a novel topoisomerase I inhibitor. J Clin Oncol. 1992 Apr;10(4):647-56. doi: 10.1200/JCO.1992.10.4.647. PMID 1312588
- [Background] Rivory LP, Robert J. [Pharmacology of camptothecin and its derivatives]. Bull Cancer. 1995 Apr;82(4):265-85. French. PMID 10846537
- [Background] Grochow LB, Rowinsky EK, Johnson R, Ludeman S, Kaufmann SH, McCabe FL, Smith BR, Hurowitz L, DeLisa A, Donehower RC, et al. Pharmacokinetics and pharmacodynamics of topotecan in patients with advanced cancer. Drug Metab Dispos. 1992 Sep-Oct;20(5):706-13. PMID 1358575
- [Background] Creemers GJ, Bolis G, Gore M, Scarfone G, Lacave AJ, Guastalla JP, Despax R, Favalli G, Kreinberg R, Van Belle S, Hudson I, Verweij J, Ten Bokkel Huinink WW. Topotecan, an active drug in the second-line treatment of epithelial ovarian cancer: results of a large European phase II study. J Clin Oncol. 1996 Dec;14(12):3056-61. doi: 10.1200/JCO.1996.14.12.3056. PMID 8955650
- [Background] Kudelka AP, Tresukosol D, Edwards CL, Freedman RS, Levenback C, Chantarawiroj P, Gonzalez de Leon C, Kim EE, Madden T, Wallin B, Hord M, Verschraegen C, Raber M, Kavanagh JJ. Phase II study of intravenous topotecan as a 5-day infusion for refractory epithelial ovarian carcinoma. J Clin Oncol. 1996 May;14(5):1552-7. doi: 10.1200/JCO.1996.14.5.1552. PMID 8622071
- [Background] ten Bokkel Huinink W, Gore M, Carmichael J, Gordon A, Malfetano J, Hudson I, Broom C, Scarabelli C, Davidson N, Spanczynski M, Bolis G, Malmstrom H, Coleman R, Fields SC, Heron JF. Topotecan versus paclitaxel for the treatment of recurrent epithelial ovarian cancer. J Clin Oncol. 1997 Jun;15(6):2183-93. doi: 10.1200/JCO.1997.15.6.2183. PMID 9196130
- [Background] Kaufmann SH, Peereboom D, Buckwalter CA, Svingen PA, Grochow LB, Donehower RC, Rowinsky EK. Cytotoxic effects of topotecan combined with various anticancer agents in human cancer cell lines. J Natl Cancer Inst. 1996 Jun 5;88(11):734-41. doi: 10.1093/jnci/88.11.734. PMID 8637027
- [Background] Rowinsky EK, Kaufmann SH, Baker SD, Grochow LB, Chen TL, Peereboom D, Bowling MK, Sartorius SE, Ettinger DS, Forastiere AA, Donehower RC. Sequences of topotecan and cisplatin: phase I, pharmacologic, and in vitro studies to examine sequence dependence. J Clin Oncol. 1996 Dec;14(12):3074-84. doi: 10.1200/JCO.1996.14.12.3074. PMID 8955652
- [Background] Miller AA, Hargis JB, Lilenbaum RC, Fields SZ, Rosner GL, Schilsky RL. Phase I study of topotecan and cisplatin in patients with advanced solid tumors: a cancer and leukemia group B study. J Clin Oncol. 1994 Dec;12(12):2743-50. doi: 10.1200/JCO.1994.12.12.2743. PMID 7527456
- [Background] O'Reilly S, Fleming GF, Barker SD, Walczak JR, Bookman MA, McGuire WP 3rd, Schilder RJ, Alvarez RD, Armstrong DK, Horowitz IR, Ozols RF, Rowinsky EK. Phase I trial and pharmacologic trial of sequences of paclitaxel and topotecan in previously treated ovarian epithelial malignancies: a Gynecologic Oncology Group study. J Clin Oncol. 1997 Jan;15(1):177-86. doi: 10.1200/JCO.1997.15.1.177. PMID 8996140
- [Background] Murren JR, Anderson S, Fedele J, Pizzorno G, Belliveau D, Zelterman D, Burtness BA, Tocino I, Flynn SD, Beidler D, Cheng YC. Dose-escalation and pharmacodynamic study of topotecan in combination with cyclophosphamide in patients with refractory cancer. J Clin Oncol. 1997 Jan;15(1):148-57. doi: 10.1200/JCO.1997.15.1.148. PMID 8996136
- [Background] Schiller JH, Kim K, Hutson P, DeVore R, Glick J, Stewart J, Johnson D. Phase II study of topotecan in patients with extensive-stage small-cell carcinoma of the lung: an Eastern Cooperative Oncology Group Trial. J Clin Oncol. 1996 Aug;14(8):2345-52. doi: 10.1200/JCO.1996.14.8.2345. PMID 8708727
- [Background] O'Reilly S, Rowinsky E, Slichenmyer W, Donehower RC, Forastiere A, Ettinger D, Chen TL, Sartorius S, Bowling K, Smith J, Brubaker A, Lubejko B, Ignacio V, Grochow LB. Phase I and pharmacologic studies of topotecan in patients with impaired hepatic function. J Natl Cancer Inst. 1996 Jun 19;88(12):817-24. doi: 10.1093/jnci/88.12.817. PMID 8637048
- [Background] Saltz L, Sirott M, Young C, Tong W, Niedzwiecki D, Tzy-Jyun Y, Tao Y, Trochanowski B, Wright P, Barbosa K, et al. Phase I clinical and pharmacology study of topotecan given daily for 5 consecutive days to patients with advanced solid tumors, with attempt at dose intensification using recombinant granulocyte colony-stimulating factor. J Natl Cancer Inst. 1993 Sep 15;85(18):1499-507. doi: 10.1093/jnci/85.18.1499. PMID 7689654
- [Background] Rowinsky EK, Grochow LB, Sartorius SE, Bowling MK, Kaufmann SH, Peereboom D, Donehower RC. Phase I and pharmacologic study of high doses of the topoisomerase I inhibitor topotecan with granulocyte colony-stimulating factor in patients with solid tumors. J Clin Oncol. 1996 Apr;14(4):1224-35. doi: 10.1200/JCO.1996.14.4.1224. PMID 8648378
- [Background] Wall JG, Burris HA 3rd, Von Hoff DD, Rodriguez G, Kneuper-Hall R, Shaffer D, O'Rourke T, Brown T, Weiss G, Clark G, et al. A phase I clinical and pharmacokinetic study of the topoisomerase I inhibitor topotecan (SK&F 104864) given as an intravenous bolus every 21 days. Anticancer Drugs. 1992 Aug;3(4):337-45. doi: 10.1097/00001813-199208000-00004. PMID 1330081
- [Background] van Warmerdam LJ, ten Bokkel Huinink WW, Rodenhuis S, Koier I, Davies BE, Rosing H, Maes RA, Beijnen JH. Phase I clinical and pharmacokinetic study of topotecan administered by a 24-hour continuous infusion. J Clin Oncol. 1995 Jul;13(7):1768-76. doi: 10.1200/JCO.1995.13.7.1768. PMID 7602366
- [Background] Rowinsky EK, Adjei A, Donehower RC, Gore SD, Jones RJ, Burke PJ, Cheng YC, Grochow LB, Kaufmann SH. Phase I and pharmacodynamic study of the topoisomerase I-inhibitor topotecan in patients with refractory acute leukemia. J Clin Oncol. 1994 Oct;12(10):2193-203. doi: 10.1200/JCO.1994.12.10.2193. PMID 7931489
- [Background] Kantarjian HM, Beran M, Ellis A, Zwelling L, O'Brien S, Cazenave L, Koller C, Rios MB, Plunkett W, Keating MJ, et al. Phase I study of Topotecan, a new topoisomerase I inhibitor, in patients with refractory or relapsed acute leukemia. Blood. 1993 Mar 1;81(5):1146-51. PMID 8382970
- [Background] Lotz JP, Pautier P, Selle F, Viens P, Fabbro M, Lokiec F, Viret F, Gligorov J, Gosse B, Provent S, Ribrag V, Miclea JM, Dosquet C, Goetschel A, Cailliot C, Lefevre G, Geneve J, Lhomme C; Groupe d' Intensification des traitements des Tumeurs Ovariennes (ITOV Group). Phase I study of high-dose topotecan with haematopoietic stem cell support in the treatment of ovarian carcinomas: the ITOV 01 protocol. Bone Marrow Transplant. 2006 Apr;37(7):669-75. doi: 10.1038/sj.bmt.1705310. PMID 16501591
- [Background] Prince HM, Rischin D, Quinn M, Allen D, Planner R, Neesham D, Gates P, Davison J. Repetitive high-dose topotecan, carboplatin, and paclitaxel with peripheral blood progenitor cell support in previously untreated ovarian cancer: results of a Phase I study. Gynecol Oncol. 2001 May;81(2):216-24. doi: 10.1006/gyno.2001.6121. PMID 11330952
- [Background] Miller AB, Hoogstraten B, Staquet M, Winkler A. Reporting results of cancer treatment. Cancer. 1981 Jan 1;47(1):207-14. doi: 10.1002/1097-0142(19810101)47:13.0.co;2-6. PMID 7459811
- [Background] Cheung YK, Chappell R. Sequential designs for phase I clinical trials with late-onset toxicities. Biometrics. 2000 Dec;56(4):1177-82. doi: 10.1111/j.0006-341x.2000.01177.x. PMID 11129476